CLINICAL TRIAL: NCT02173821
Title: A Follow-up Study to Examine the Presence of Anti-human Growth Hormone Antibodies Following a Randomised, Open-label, Parallel-group, Multi-centre Trial (FE 999905 CS07) in Which the Efficacy and Safety of 12 Months' Treatment With One Daily Dose of ZOMACTON Were Compared to One Daily Dose of GENOTROPIN
Brief Title: A Follow-up Study to Examine the Presence of Anti-human Growth Hormone Antibodies Following a Study (FE 999905 CS07) of Zomacton in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000134; 2014-000627-24 (EudraCT Number)
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Idiopathic Growth Hormone Deficiency
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling — Blood sample will be collected at a single visit

SUMMARY:
This is a follow-up study of patients, treated with one daily dose of Zomacton or one daily dose of Genotropin in the previously completed FE 999905 CS07 trial, who had presence of anti-hGH antibodies at any post-dosing visit during the 12-month treatment period. No investigational medicinal product will be administered in connection with this follow-up study. Eligible patients will attend one visit in this follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in trial FE 999905 CS07 and presence of anti-hGH antibodies at any post-dosing visit throughout the 12-month treatment period
* Signed informed consent and obtained assent according to local rules and practice
* Information on medical history, concomitant medications, and growth hormone therapy since completion of trial FE 999905 CS07

Exclusion Criteria:

* There are no pre-defined exclusion criteria in this study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of anti-human Growth Hormone (hGH) antibodies | At visit 1
  Measured as percentage of patients with positive anti-hGH antibodies.

SECONDARY OUTCOMES:
Prevalence of neutralising antibodies in confirmed positive anti-hGH antibody samples | At visit 1
  Measured as percentage of patients with neutralising antibodies in patients with confirmed positive anti-hGH antibody samples.
Binding capacity levels in confirmed anti-hGH antibody positive samples | At visit 1
  Measured as percentage of patients with binding capacity <2 mg/L in patients with confirmed positive anti-hGH antibody samples.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (7):
- Szent János Kórház és Észak Budai Egyesített Kórházai (there may be other sites in this country), Budapest, Hungary
- Seth GSMC & KEM Hospital (there may be other sites in this country), Maharashtra, India
- The Chaim Sheba Medical Center (there may be other sites in this country), Ramat Gan, Israel
- Uniwersyteckie Centrum Kliniczne (there may be other sites in this country), Gdansk, Poland
- Paediatric Endocrinology/Medicali's SRL (there may be other sites in this country), Timișoara, Romania
- Federal State Institution "Endocrinology Scientific Center of Rosmedtechnology" (there may be other sites in this country), Moscow, Russia
- Institute of Endocrinology and Metabolism named after Komisarenko of AMS Ukraine (there may be other sites in this country), Kiev, Ukraine